CLINICAL TRIAL: NCT04303208
Title: Sirtuin 3 and Sirtuin 7 in Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mai Hany Ahmed Ibrahim, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SIRT 3 and SIRT 7 in SSC
Record Dates: First submitted 2020-03-03; First posted 2020-03-11 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Other): Blood sample ( 5 ml venous blood ) will be obtained under complete aseptic conditions from all eligible participants , using serum separator tube and allow samples to clot for 30 minutes before centrifugation for 15 minutes to obtain clear serum .Separated serum will be stored at < - 20c ( avoid repeated freeze - thaw cycles) till assessment of Sirt 3 and Sirt 7 levels using Enzyme- linked immunosorbent assay (ELISA) method .
  Interventions: Procedure: Blood sample
- control group (Other): Blood sample ( 5 ml venous blood ) will be obtained under complete aseptic conditions from all eligible participants , using serum separator tube and allow samples to clot for 30 minutes before centrifugation for 15 minutes to obtain clear serum .Separated serum will be stored at < - 20c ( avoid repeated freeze - thaw cycles) till assessment of Sirt 3 and Sirt 7 levels using Enzyme- linked immunosorbent assay (ELISA) method .
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Blood sample ( 5 ml venous blood ) will be obtained under complete aseptic conditions from all eligible participants , using serum separator tube and allow samples to clot for 30 minutes before centrifugation for 15 minutes to obtain clear serum . Separated serum will be stored at < - 20c ( avoid repeated freeze - thaw cycles ) till assessment of Sirt 3 and Sirt 7 levels using Enzyme- linked immunosorbent assay (ELISA) method .

SUMMARY:
Systemic sclerosis (SSc) is a systemic autoimmune disease in which inflammation and fibrosis play a crucial role and lead to severe damage and failure of multiple organs such as the skin, joints, tendons, gastrointestinal tract, lungs, heart, blood vessels, and kidneys. It primarily affects women but disease is often more severe in males.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a systemic autoimmune disease in which inflammation and fibrosis play a crucial role and lead to severe damage and failure of multiple organs such as the skin, joints, tendons, gastrointestinal tract, lungs, heart, blood vessels, and kidneys. It primarily affects women but disease is often more severe in males.

Sirtuins are a class of nicotinamide adenine dinucleotide-consuming enzymes that are implicated in numerous biological pathways .

Sirtuins are considered among the most promising targets for modulating aging-associated cellular and molecular processes and disease pathologies , The majority of studies have shown decreased SIRT expression in tissues and fibroblasts from patients with SSc compared to controls and in experimental fibrosis in mice .

Decreased SIRT3 levels and activity were observed in fibrotic areas of SSc and IPF lung tissues and SSc skin biopsies and explanted fibroblasts compared to controls , Wyman et al investigated the expression of all seven mammalian SIRTs in lung tissues and fibroblasts from patients with SSc and IPF and found a tendency for SIRTs to be decreased in patients with fibrosis compared to controls , with a particularly notable decline in SIRT7 .

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis diagnosed by 2013 ACR\EULAR classification criteria of systemic sclerosis
* Patients' age >18
* 25 rheumatoid arthritis patients as a control .

Exclusion Criteria:

-Overlap or mixed connective tissue diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
: To measure circulating Sirt 3 and Sirt 7 levels in patients with systemic sclerosis and their relation with different clinical manifestations | 2 years
  the amount of Sirt 3 and Sirt 7 will be measured by ELISA
Influence of Sirt 3 and Sirt 7 in fibrosis in Systemic sclerosis | 2 years
  the amount of Sirt 3 and Sirt 7 will be measured by ELISA